CLINICAL TRIAL: NCT04750213
Title: Post-marketing Observational Study for Humira in Participants Diagnosed With Pyoderma Gangrenosum (PG)
Brief Title: A Study to Assess Adverse Events and Change in Disease State in Adult Participants Being Treated With Humira in Participants Diagnosed With Pyoderma Gangrenosum (PG)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-251
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pyoderma Gangrenosum
Keywords: Pyoderma Gangrenosum; Humira; Adalimumab
MeSH Terms: conditions — Pyoderma Gangrenosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Humira (Adalimumab): Participants receiving Adalimumab for Pyoderma Gangrenosum (PG).

SUMMARY:
Pyoderma Gangrenosum (PG) is a rapidly progressive disease and presents as painful, single or multiple lesions, with several clinical variants, in different locations, with a nonspecific histology, which makes the diagnosis challenging and often delayed. The main objective of this study is to estimate the incidence proportion of all the infection reported as adverse drug reaction (ADR) of Humira with PG participants.

Humira is the only drug approved for the treatment of Pyoderma Gangrenosum (PG) in Japan. Approximately 60 adult participants with PG at approximately 60 sites in Japan.

Participants will receive injectable Humira (Adalimumab) as prescribed by the physician prior to enrolling in this study.

There may be a higher burden for participants in this study compared to standard of care. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and by verbal interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Pyoderma Gangrenosum (PG).
* Have been prescribed Humira for PG treatment within 14 days.

Exclusion Criteria:

- Have Pyoderma Gangrenosum (PG) in previous treatment with Humira.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence Percentage of all the Infection Reported as Adverse Drug Reaction (ADR) | Up to 52 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.

SECONDARY OUTCOMES:
Incidence Percentage of Serious Infection Reported as ADR | Up to 52 weeks
  An AE is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.
Incidence Percentage of each ADR (Besides Infection) | Up to 52 weeks
  An AE is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment. Among AEs, an event whose causal relationship with the product cannot be ruled out is considered an adverse drug reaction.
Change in Physician's Global Assessment (PGA) [Global] Grade | Up to Week 52
  PGA will be used for overall assessment of efficacy.
Change in PGA [Target] Grade | Up to Week 52
  PGA will be used for assessment of efficacy of target lesions.
Change in Investigator Inflammation Assessment (IIA) Score from Start of Dosing | Up to Week 52
  IIA will be used for assessment of efficacy of target lesions.
Change in Verbal Rating Scale (VRS) Category | Up to Week 52
  Pain improvement will be assessed using a VRS scale 0-3 with a lower score indicating less pain.
Percentage of Participants with Recurrence | Up to Week 52
  Recurrence of PG.
Time to Recurrence (Day) | Up to Week 52
  Recurrence of PG.
Percentage of PG Subtype at Recurrence | Up to Week 52
  Recurrence of PG. PG subtypes include (ulcerative (including peristomal), bullous, pustular, vegetative).
Pain Improvement Assessed with VRS | Week 26 to Week 52
  Pain improvement will be assessed using a VRS scale 0-3 with a lower score indicating less pain.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (46):
- Japan (46):
  - NHO Nagoya Medical Center /ID# 246013, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 233778, Nagoya, Aichi-ken
  - Akita University Hospital /ID# 242706, Akita, Akita
  - Kyushu University Hospital /ID# 247492, Fukuoka, Fukuoka
  - Japanese Red Cross Fukuoka Hospital /ID# 244051, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 246502, Kurume-shi, Fukuoka
  - Central Japan International Medical Center /ID# 239391, Minokamo-shi, Gifu
  - Gunma University Hospital /ID# 239390, Maebashi, Gunma
  - Sapporo Medical University Hospital /ID# 241180, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 252567, Sapporo, Hokkaido
  - Hokkaido Medical Center /ID# 251657, Sapporo, Hokkaido
  - Kansai Rosai Hospital /ID# 246592, Amagasaki-shi, Hyōgo
  - Kobe University Hospital /ID# 249396, Kobe, Hyōgo
  - Nishi-Kobe Medical Center /ID# 244224, Kobe, Hyōgo
  - Ishikawa Prefectural Central Hospital /ID# 239089, Kanazawa, Ishikawa-ken
  - Kanazawa University Hospital /ID# 248730, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital /ID# 240576, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital /ID# 250193, Takamatsu, Kagawa-ken
  - Teikyo University Mizonokuchi Hospital /ID# 244693, Kawasaki, Kanagawa
  - Yokohama Municipal Citizen's Hospital /ID# 233779, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hosp /ID# 252892, Yokohama, Kanagawa
  - Kumamoto University Hospital /ID# 244050, Kumamoto, Kumamoto
  - Fukuchiyama City Hospital /ID# 246593, Fukuchiyama-shi, Kyoto
  - Mie University Hospital /ID# 238747, Tsu, Mie-ken
  - Tohoku University Hospital /ID# 252113, Sendai, Miyagi
  - Tohoku Medical and Pharmaceuti /ID# 230270, Sendai, Miyagi
  - University of Miyazaki Hospital /ID# 241179, Miyazaki, Miyazaki
  - Shinshu University Hospital /ID# 230272, Matsumoto-shi, Nagano
  - Nara Medical University Hospital /ID# 241880, Kashihara-shi, Nara
  - Okayama University Hospital /ID# 238746, Okayama, Okayama-ken
  - Okinawa Kyodo Hospital /ID# 241739, Naha, Okinawa
  - Naha City Hospital /ID# 240818, Naha, Okinawa
  - University of the Ryukyus Hospital /ID# 252114, Nakagami-gun, Okinawa
  - Kansai Medical University Hospital /ID# 228783, Hirakata-shi, Osaka
  - Japanese Red Cross Osaka Hospital /ID# 228782, Osaka, Osaka
  - Kindai University Hospital /ID# 252568, Osakasayama-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center /ID# 248731, Koshigaya, Saitama
  - Hamamatsu University Hospital /ID# 240817, Hamamatsu, Shizuoka
  - Chutoen General Medical Center /Id# 228780, Kakegawa-shi, Shizuoka
  - Shizuoka Saiseikai Genaral Hospital /ID# 239088, Shizuoka, Shizuoka
  - The University of Tokyo Hospital /ID# 250194, Bunkyo-ku, Tokyo
  - The Jikei University Hospital /ID# 252112, Minato-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 233780, Shinjuku-ku, Tokyo
  - Yamanashi Kosei Hospital /ID# 242168, Yamanashi, Yamanashi
  - Takatsuki General Hospital /ID# 244694, Osaka
  - Teikyo University Hospital /ID# 239389, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com